CLINICAL TRIAL: NCT06775691
Title: Comparison of Upper Extremity Function, Physical Activity Levels and Peripheral Muscle Strength, Fear of Movement, Balance, Activities of Daily Living and Quality of Life in Patients With Pacemakers According to Pacemaker Type
Status: Recruiting | Type: Observational
Sponsor: Erol Olcok Corum Training and Research Hospital (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gamze Nur AHISKALI, Physiotherapist Gamze Nur AHISKALI, Erol Olcok Corum Training and Research Hospital
Other Study IDs: 2024-08/1
Record Dates: First submitted 2024-09-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Pacemaker; Implantable Cardioverter Defibrillator; Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Pacemaker - PM
- Group 2: Implantable Cardioverter Defibrillator - ICD
- Group 3: Cardiac Resynchronization Therapy - CRT

SUMMARY:
While research and clinical practice have demonstrated the objective benefits of pacemaker use on mortality, morbidity, and quality of life, some patients do not experience the expected level of improvement following device implantation. The purpose of this research was to determine the effects of device implantation on daily living activities, upper extremity functions, peripheral muscle strength, balance problems, fear of movement and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 months have passed since pacemaker implantation and there are no complications in the last pacemaker control,
* Being in NYHA class I-II-III,
* Patients with no coordination problems,
* Volunteering to participate in the research

Exclusion Criteria:

* Patients with a history of shoulder pathologies prior to pacemaker implantation that may restrict movement of the upper limb (conditions such as severe pain around the shoulder, edema or shoulder dislocation that may restrict upper limb movement),
* Patients with a history of shoulder surgery (limitation in range of motion),
* Patients who have had a cerebrovascular event resulting in mastectomy or arm involvement on the affected side,
* Patients with decompensated heart failure,
* Patients with a history of ICD inappropriate shock,
* Those with acute myocardial infarction,
* Patients with malignancy on active treatment, patients with collagen tissue disease receiving systemic steroids,
* Chronic kidney disease patients on dialysis with unstable volume load

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who regularly visit for pacemaker check-ups will be invited to participate in the study.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of upper extremity functional capacity | 1 years
  6 Minute Peg Board ve Ring Testi - 6PBRT
Evaluation of peripheral muscle strength | 1 years
  Jamar Hydraulic Hand Dynamometer (Baseline Hydraulic Hand Dynamometer, Model: 12-0240, Fabrication Enterprises INC. White Plains, NY 10602 U.S.A.)
Evaluation of balance | 1 years
  Time Up and Go Test - TUG
Evaluation of fear of movement | 1 years
  Tampa Scale of Kinesiophobia for Heart- TSK- HEART / The person receives a total score between 17 and 68. A high score on the scale indicates a high level of kinesiophobia.
Evaluation of physical activity levels | 1 years
  International Pyhsical Activity Questionnaire Short Form, IPAQ / It is calculated using the metabolic equivalent method (MET). There are three different categories. The first category is inactive (<600 MET-minute/week), the second category is minimally active (600-300 MET-minute/week) and the last category is always active (<3000 MET-minute/week).
Evaluation of activities of daily living | 1 years
  Performance Measure for Activities of Daily Living-8 for Patient with Mild Symptomatic Heart Failure- PMADL-8 / The total score ranges from 8-32, with a high score indicating a level of limitation in activities of daily living.
Evaluation of quality of life | 1 years
  Short Form- 36 -SF-36 / Each sub-parameter is scored between 0 and 100. A high score indicates that the individual has a high quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Hitit University Corum Erol Olçok Training and Research Hospital, Çorum, Center, Turkey (Türkiye)